CLINICAL TRIAL: NCT00284050
Title: A Randomized, Double-masked, Multi-center, Phase II Study Assessing the Safety and Efficacy of Two Concentrations of Ranibizumab (Intravitreal Injections) Compared With Non-treatment Control for the Treatment of Diabetic Macular Edema With Center Involvement
Brief Title: Safety and Efficacy of Ranibizumab in Diabetic Macular Edema With Center Involvement
Acronym: RESOLVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRFB002D2201
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Results first posted 2011-01-20 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Diabetic Macular Edema
Keywords: DME; Diabetic macular edema; ranibizumab; Diabetic macular edema with center involvement
MeSH Terms: interventions — Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (3):
- Ranibizumab 0.3 mg (Experimental): Participants received monthly intravitreal injections with 0.3 mg ranibizumab (6 mg/ml) for up to 12 months. At each monthly visit from month 1 and onwards, the evaluating physician decided whether an increase in the dose to 0.6 mg was needed according to set criteria. If the dose was increased, all subsequent administrations were of the higher dose unless treatment had been withheld for more than 45 days (for any reason), in which case injections restarted with the initial dose. Laser photocoagulation was permitted as rescue treatment for the study eye after 3 consecutive monthly injections.
  Interventions: Drug: Ranibizumab 0.3 mg
- Ranibizumab 0.5 mg (Experimental): Participants received monthly intravitreal injections with 0.5 mg ranibizumab (10 mg/ml) for up to 12 months. At each monthly visit from month 1 and onwards, the evaluating physician decided whether an increase in the dose to 1.0 mg was needed according to set criteria. If the dose was increased, all subsequent administrations were of the higher dose unless treatment had been withheld for more than 45 days (for any reason), in which case injections restarted with the initial dose. Laser photocoagulation was permitted as rescue treatment for the study eye after 3 consecutive monthly injections.
  Interventions: Drug: Ranibizumab 0.5 mg
- Sham injection (Sham Comparator): Participants in the control group received 12 monthly sham intravitreal injections. The evaluation was performed using the same criteria for dose doubling as in active treatment groups. The injection was a mimicked by an empty syringe without a needle. Laser photocoagulation was permitted as rescue treatment for the study eye after 3 consecutive monthly injections.
  Interventions: Drug: Sham injection

INTERVENTIONS:
Drug: Ranibizumab 0.3 mg — 6 mg/ml ranibizumab solution for intravitreal injection
  Arms: Ranibizumab 0.3 mg
Drug: Ranibizumab 0.5 mg — 10 mg/ml ranibizumab solution for intravitreal injection
  Arms: Ranibizumab 0.5 mg
Drug: Sham injection — Non-treatment control for sham intravitreal injection.
  Arms: Sham injection

SUMMARY:
This study evaluated the safety and efficacy of ranibizumab on retinal edema and visual acuity in patients with diabetic macular edema with center involvement.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic macular edema with center involvement in at least one eye
* Type 1 or type 2 diabetes mellitus diagnosed 2 years prior to screening
* Laser photocoagulation in the study eye can be withheld for at least 3 months after randomization

Exclusion Criteria:

* Patients with uncontrolled systemic or ocular diseases
* Have any history of any intraocular surgery in the study eye within the past 6 months preceding screening
* Conditions that require chronic concomitant therapy with systemic or topical ocular corticosteroids

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis, Basel, Switzerland

REFERENCES:
- [Derived] Massin P, Bandello F, Garweg JG, Hansen LL, Harding SP, Larsen M, Mitchell P, Sharp D, Wolf-Schnurrbusch UE, Gekkieva M, Weichselberger A, Wolf S. Safety and efficacy of ranibizumab in diabetic macular edema (RESOLVE Study): a 12-month, randomized, controlled, double-masked, multicenter phase II study. Diabetes Care. 2010 Nov;33(11):2399-405. doi: 10.2337/dc10-0493. PMID 20980427

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection
Started | 51 | 51 | 49
Completed | 46 | 46 | 40
Not Completed | 5 | 5 | 9
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Lack of Efficacy | 0 | 1 | 3
Not completed — Protocol Violation | 0 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 2 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection | Total
Number analyzed (Participants) | 51 | 51 | 49 | 151
Age Continuous [Mean (Standard Deviation); unit: years] | 63.2 (10.44) | 62.8 (10.14) | 65.0 (9.26) | 63.6 (9.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 24 | 70
  Male | 29 | 27 | 25 | 81

OUTCOME MEASURES:

1. Primary Outcome: Difference Between the Baseline Level of Visual Acuity (Letters) of the Study Eye and the Mean Visual Acuity Averaged Over All Monthly Post-baseline Assessments From Month 1 to Month 12
Description: Visual acuity (VA) was assessed on both eyes during every study visit using best correction determined from protocol refraction. VA measurements were performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a testing distance of 4 meters as described in the Study Operations Manual.
Time Frame: Baseline through the end of study (Month 12)
Population: Full Analysis Set (FAS): All patients who received at least one application of study treatment and had at least one post-baseline assessment for BCVA. A Last Observation Carried Forward (LOCF) approach was used; missing values were replaced by the mean of the last observation before and the first observation after the missing time-point.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 51 | 51 | 49
Letters | 9.2 (5.60) | 6.4 (9.21) | -0.1 (9.77)

2. Primary Outcome: Mean Change From Baseline in Visual Acuity (Letters) of the Study Eye at Month 12
Description: as for outcome 1
Time Frame: Baseline through the end of study (Month 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 51 | 51 | 49
Letters | 11.8 (6.59) | 8.8 (10.99) | -1.4 (14.16)

3. Secondary Outcome: Mean Change From Baseline in Central Retinal Thickness (µm) of the Study Eye at Month 12
Description: Optical Coherence Tomography (OCT) was assessed on both eyes at every study visit. These assessments were performed by trained personnel at the sites. OCT imaging was performed using the Zeiss Humphrey System Model 2000 (or later) with version A6.1 software running under Windows 95 or Windows 98. The analysis of the OCT images were performed by the Photographic Reading Center which provided a study manual and training materials. OCT operators, systems and software were certified prior to any evaluation of study patients.
Time Frame: Baseline through the end of study (Month 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 51 | 51 | 49
µm | -200.7 (122.18) | -187.6 (147.82) | -48.4 (153.43)

ADVERSE EVENTS:
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection
Serious Adverse Events (participants affected / at risk) | 9/51 | 9/51 | 9/49
Other Adverse Events (participants affected / at risk) | 37/51 | 43/51 | 32/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.3 mg (N=51) | Ranibizumab 0.5 mg (N=51) | Sham Injection (N=49)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Endophthalmitis (Study eye) (Eye disorders) | 1 | 1 | 0
Retinal artery occlusion (Study eye) (Eye disorders) | 0 | 1 | 0
Retinal detachment (Study eye) (Eye disorders) | 0 | 0 | 1
Retinal ischaemia (Study eye) (Eye disorders) | 0 | 1 | 0
Vitreous haemorrhage (Study eye) (Eye disorders) | 1 | 0 | 0
Pitting oedema (General disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Diabetic gangrene (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Infected epidermal cyst (Infections and infestations) | 0 | 1 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.3 mg (N=51) | Ranibizumab 0.5 mg (N=51) | Sham Injection (N=49)
Cataract (Fellow eye) (Eye disorders) | 0 | 4 | 2
Conjunctival haemorrhage (Study eye) (Eye disorders) | 10 | 13 | 7
Conjunctival hyperaemia (Study eye) (Eye disorders) | 2 | 1 | 3
Conjunctivitis (Fellow eye) (Eye disorders) | 1 | 0 | 4
Conjunctivitis (Study eye) (Eye disorders) | 1 | 1 | 4
Corneal disorder (Study eye) (Eye disorders) | 3 | 2 | 0
Eye irritation (Study eye) (Eye disorders) | 3 | 1 | 1
Eye pain (Study eye) (Eye disorders) | 9 | 9 | 10
Eye pruritus (Study eye) (Eye disorders) | 3 | 2 | 2
Eyelid oedema (Study eye) (Eye disorders) | 1 | 0 | 3
Foreign body sensation in eyes (Study eye) (Eye disorders) | 3 | 3 | 1
Lacrimation increased (Study eye) (Eye disorders) | 4 | 4 | 0
Macular oedema (Fellow eye) (Eye disorders) | 3 | 2 | 0
Ocular hyperaemia (Study eye) (Eye disorders) | 2 | 2 | 4
Retinal disorder (Study eye) (Eye disorders) | 3 | 1 | 0
Retinal exudates (Study eye) (Eye disorders) | 2 | 1 | 4
Retinal haemorrhage (Study eye) (Eye disorders) | 1 | 2 | 3
Visual acuity reduced (Study eye) (Eye disorders) | 1 | 6 | 5
Visual disturbance (Study eye) (Eye disorders) | 3 | 1 | 1
Vitreous floaters (Study eye) (Eye disorders) | 1 | 8 | 0
Vitreous haemorrhage (Fellow eye) (Eye disorders) | 3 | 4 | 3
Vitreous haemorrhage (Study eye) (Eye disorders) | 0 | 4 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 3
Bronchitis (Infections and infestations) | 1 | 3 | 2
Influenza (Infections and infestations) | 2 | 3 | 1
Nasopharyngitis (Infections and infestations) | 5 | 5 | 1
Intraocular pressure increased (Fellow eye) (Investigations) | 1 | 3 | 0
Intraocular pressure increased (Study eye) (Investigations) | 6 | 15 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
Hypertension (Vascular disorders) | 3 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.